CLINICAL TRIAL: NCT04754659
Title: Renal Function After Stentgraft Treatment Of Abdominal Aneurysm With Supra- Versus Infrarenal Fixation - a Randomized Clinical Study
Brief Title: Renal Function After Stentgraft Treatment Of Abdominal Aortic Aneurysm
Acronym: RENOFIX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RENOFIX 3.1
Record Dates: First submitted 2021-01-12; First posted 2021-02-15 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Aortic Aneurysm, Abdominal; Renal Insufficiency; Stent-Graft Thrombosis
Keywords: abdominal aortic aneurysm; postoperative renal failure; stentgraft complication
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Renal Insufficiency

STUDY DESIGN:
Intervention Model Description: Randomized controlled, parallel group, partly blinded clinical study.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The type of stentgraft is masked for participants, investigators and outcome assessors as the journal chart and information about implanted device are made not accessible for the above mentioned individuals, and all data will be gathered in an Electronic Case Report Form (eCRF) with stentgraft information masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Suprarenal (Experimental): Individuals that are treated with a suprarenal stentgraft for a previously diagnosed AAA.
  Interventions: Device: Stentgraft
- Infrarenal (Active Comparator): Individuals that are treated with an infrarenal stentgraft for a previously diagnosed AAA.
  Interventions: Device: Stentgraft

INTERVENTIONS:
Device: Stentgraft — Stentgraft treatment for AAA. Comparison between supra vs infrarenal fixation.

SUMMARY:
This randomized controlled trial aim to determine the impact on renal function after treatment for infrarenal abdominal aortic aneurysm (AAA) with stentgrafts either with active supra- or infrarenal fixation.

DETAILED DESCRIPTION:
This randomized controlled trial aim to determine the impact on renal function after treatment for infrarenal abdominal aortic aneurysm with stentgrafts either with active supra- or infrarenal fixation. Individuals are planned to be included throughout Scandinavia. After inclusion in the study, baseline data is collected and computerized randomization between the two stent graft fixation types is performed. Follow-up will be scheduled after 1 month and 1,3 and 5 years. Analyses of blood samples to determine renal function are undertaken together with CT scans to detect stentgraft performance at all follow-up visits alongside assessments of health-related quality of life questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent
* Meet criteria for non-ruptured infrarenal/iliac aneurysm
* Suitable anatomy for treatment with an approved device (CE-marked) stentgraft according to the manufacturers' instructions for use for AAA.
* Accepted for treatment with endovascular aortic repair (EVAR) by the participating vascular center.

Exclusion Criteria:

* Ongoing or planned dialysis
* AAA treatment requiring stents or stentgrafts in renal and/or visceral arteries
* Inability to independently complete HRQoL questionnaires due to language barriers
* Anatomical preconditions that do not allow both types of fixation to be used interchangeably, i.e. very advanced suprarenal tortuosity (>60 degrees), advanced suprarenal dilatation or infrarenal thrombus >25% of circumference.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2022-12-19 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with decreased renal function (composite endpoint together with the endpoint below) | Change between baseline renal function and at 3 years.
  Decrease of more than 20 percent in estimated Glomerular Filtration Rate (eGFR) after stentgraft treatment.
Number of participants with new renal infarct | Change in numbers of new renal infarcts between baseline and at 3 years.
  Diagnosed new renal infarct on CT scan after treatment

SECONDARY OUTCOMES:
Number of participants with decreased renal function and new renal infarct (Analysis of the individual components of the primary composite endpoint at 1, 3 and 5 years). | From treatment and 1, 3 and 5 years postoperatively
  Analysis of individual endpoints (decrease of more than 20 percent in estimated Glomerular Filtration Rate (eGFR) after stentgraft treatment and diagnosed new renal infarct on CT scan after treatment).
Number of participants with decreased score in quality of life-questionnaire | From treatment and 1 and 3 years postoperatively
  Change in life quality questionnaire (Research and development questionnaire 36 (RAND-36)) one and three years after surgery compared with baseline data collected prior to surgery. Score in the scale are between 0 and 100 and decreased score indicate worse outcome.
Number of participants with stentgraft thrombosis | From treatment and 1, 3 and 5 years postoperatively
  Occurence of stentgraft thrombosis postoperatively at 1 month, 1, 3 and 5 years.
Number of participants with aneurysm related mortality | From treatment and 1, 3 and 5 years postoperatively
  Aneurysm related mortality postoperatively at 1 month, 1, 3 and 5 years.
Number of participants with aneurysm related hospitalizations | From treatment and 1, 3 and 5 years postoperatively
  Aneurysm related hospitalizations postoperatively at 1 month, 1, 3 and 5 years.
Number of participants with continuing aneurysm growth | From treatment and 1, 3 and 5 years postoperatively
  Continuing aneurysm growth postoperatively at 1 month, 1, 3 and 5 years.
Number of participants with new diagnosis of cancer | From treatment and 1, 3 and 5 years postoperatively
  New diagnosis of cancer postoperatively at 1 month, 1, 3 and 5 years.

OTHER OUTCOMES:
Number of participants with migration (Safety endpoint composite together with the endpoints below) | From treatment and 1, 3 and 5 years postoperatively
  Migration (stentgraft migration more than 3mm) postoperatively at 1 month, 1, 3 and 5 years.
Number of participants with diagnosed endoleak | From treatment and 1, 3 and 5 years postoperatively
  Re-intervention for endoleak postoperatively at 1 month, 1, 3 and 5 years.
Number of participants with aortic rupture | From treatment and 1, 3 and 5 years postoperatively
  Occurence of postoperative aortic rupture postoperatively at 1 month, 1, 3 and 5 years.
Number of participants with renal artery thrombosis | From treatment and 1, 3 and 5 years postoperatively
  Postoperative renal artery thrombosis postoperatively at 1 month, 1, 3 and 5 years.
Number of participants with renal artery stenosis | From treatment and 1, 3 and 5 years postoperatively
  Occurence of postoperative renal artery stenosis postoperatively at 1 month, 1, 3 and 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Lindgren, M.D, Study Chair — Department of Hybrid and Interventional Surgery, Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, VastraGotaland, Sweden

IPD SHARING:
Plan to Share IPD: No